CLINICAL TRIAL: NCT06615492
Title: RoutinE Versus On-demand Intraoperative Extracorporeal Membrane Oxygenation (ECMO) During LUng TransplantatION (REVOLUTION)
Brief Title: Routine vs On-demand ECMO for Lung Transplantation
Acronym: REVOLUTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-11391
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Failure; Interstitial Lung Disease (ILD); Pulmonary Fibrosis; COPD (Chronic Obstructive Pulmonary Disease)
Keywords: ECMO; Lung Transplantation
MeSH Terms: conditions — Respiratory Insufficiency; Lung Diseases, Interstitial; Pulmonary Fibrosis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine ECMO (Experimental): Routine ECMO during lung tansplant
  Interventions: Device: Routine ECMO
- On-demand ECMO (Active Comparator): Selective, indication-based intraoperative cardiopulmonary support.
  Interventions: Device: On-demand ECMO

INTERVENTIONS:
Device: Routine ECMO — Routine intraoperative venoarterial ECMO during lung transplant
  Arms: Routine ECMO
Device: On-demand ECMO — Selective, indication-based intraoperative cardiopulmonary support. In this group, the transplant will be planned without cardiopulmonary support. intraoperative venoarterial ECMO will be used selectively based on hemodynamic and/or gas exchange abnormalities :
  1. Inability to maintain adequate hemodynamics and stable perfusion despite volume resuscitation and vasopressor administration and in the absence of readily correctable cause
  2. Inability to tolerate pulmonary artery clamping
  3. Inadequate gas exchange despite attempts at the optimization of ventilator parameters and treatments related to respiratory mechanics and ventilation/perfusion matching
  4. Inadequate exposure to the surgical field
  5. The transplant team is concerned about the ability to maintain organ perfusion or ventilate with a lung protective strategy, even if the aforementioned criteria are unmet.
  6. Concerns about donor lung quality and a desire to protect the implanted lung from single lung perfusion
  Arms: On-demand ECMO

SUMMARY:
Lung transplantation is a complex procedure performed in patients with terminal lung disease. The transplant procedure stresses the patient's heart and lungs, which are already taxed by the underlying disease process. The heart-lung machine is occasionally used to support the patient and ensure adequate oxygen supply to other organs during the operation. It can be used routinely in all patients or selectively in patients who exhibit reduced oxygen supply to the remaining organs. This process, known as cardiopulmonary bypass (CPB), pumps blood out of the body to a heart-lung machine that removes carbon dioxide and returns oxygen-filled blood to the body.

Although using the CPB increases the risk of bleeding, infection, and coagulation complications, it should still be considered in high-risk patients to compensate for more severe complications such as kidney failure and stroke caused by a lack of cardiopulmonary support. Extracorporeal membrane oxygenation (ECMO) is a recently developed CPB variation associated with fewer bleeding complications. It has recently replaced the traditional heart-lung machine as the preferred method of cardiopulmonary support during lung transplantation. Since ECMO is associated with fewer complications than standard CPB, many centers have increased their use of ECMO during lung transplantation. Some have even employed it routinely. However, there remains significant debate on how often it should be used.

Therefore, the study's main objective is to compare the two approaches in lung transplantation, i.e., routine use versus selective use, and to determine if one approach is preferable to the other.

DETAILED DESCRIPTION:
This study compares two approaches to intraoperative cardiopulmonary support during lung transplantation: routine cardiopulmonary support with extracorporeal membrane oxygenation (ECMO) versus selective use. Despite recent improvements in lung transplant outcomes, postoperative complications are common. Intraoperative hemodynamic management is vital to the success of lung transplantation. Many centers, including all four Canadian centers, use ECMO to provide intraoperative support. However, lung transplantation without cardiopulmonary support may be possible in certain patients. In such patients, the transplant may be started without ECMO. ECMO may be initiated "on-demand" if hemodynamic embarrassment or hypoxia occurs. Conversely, the opposite approach would be routinely conducting all lung transplants using ECMO. The current practice in many centers is to use ECMO selectively. By extension, the investigators believe that more liberal use of intraoperative ECMO will produce less intraoperative hemodynamic instability and hypoxia. However, it is unclear the extent of ECMO use necessary to improve the incidence of postoperative hypoperfusion-related complications. Should ECMO be used routinely in all patients or selectively based on the intraoperative course? The study is a prospective, randomized, controlled trial with two treatment arms: routine support with ECMO versus selective (on-demand) support with ECMO. Study population (Inclusion and exclusion criteria): All patients, 18 years of age or older, undergoing lung transplantation will be screened for participation. We will exclude patients who require intraoperative ECMO, multi-organ transplants, and retransplantation Arms and Interventions: On-demand ECMO: The transplant will be planned without cardiopulmonary support in this group. Intraoperative ECMO will be employed if there is an inability to maintain adequate organ perfusion and oxygen delivery despite resuscitation. Routine ECMO: Routine intraoperative ECMO in all patients, regardless of hemodynamic status. Primary outcome: Intensive care unit (ICU)-free days in the first 28 days post-lung transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lung transplant surgery

Exclusion Criteria:

* Inability to provide consent for the study
* Retransplantation
* Multi-organ transplantation
* Contra-indication to standard heparin anticoagulation (e.g., heparin-induced thrombocytopenia)
* Lung transplant recipients where intraoperative cardiopulmonary support is mandatory:
* Severe pulmonary hypertension (PH):

  1. Systolic pulmonary artery pressure (PAP) ≥ 80 mm Hg on the most recent echocardiography, right heart catheterization, or pulmonary artery catheter measurement
  2. Mean PAP ≥ 55 mm Hg on the most recent echocardiography, right heart catheterization, or pulmonary artery catheter measurement
  3. The ratio of mean pulmonary to systemic artery pressure of > 0.66
* Moderate to severe right ventricular (RV) hypokinesis or dysfunction
* Left ventricular dysfunction: Defined as ejection fraction (LVEF) less than 45% on echocardiography, ventriculography, computed tomography (CT), or magnetic resonance imaging (MRI)
* Patients requiring concomitant cardiac surgery: For example, significant coronary artery disease (CAD) requiring surgical grafting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2028-11-05 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
ICU-free days | From the end of surgery up to 28 days after surgery
  Intensive care unit (ICU)-free days in the first 28 days post-lung transplant (28 minus the ICU length of stay)

SECONDARY OUTCOMES:
Incidence and grade of primary graft dysfunction (PGD) at 0, 24, 48, and 72 hours | From the end of surgery up to 72 hours after surgery
  The definition is based on the criteria for the International Society of Heart and Lung Transplantation (ISHLT) grading system.
Incidence of all-cause mortality | From the end of surgery to 90 days after surgery
  Death, whatever the cause
Incidence of intraoperative blood product transfusion requirements | Beginning from the surgical incision up to the arrival to the intensive care unit immediately after surgery
  Number of packed red blood cell units and total blood product units (red blood cells, plasma, platelets, prothrombin complex concentrates) transfused.
Incidence of perioperative blood product transfusion | From the beginning of surgery up to 72 hours after surgery.
  Number of packed red blood cell units and total blood product units (red blood cells, plasma, platelets, prothrombin complex concentrates) transfused.
Intensive care unit and hospital length of stay in days | Beginning from the arrival to the intensive care unit immediately after surgery
  Lenght of stay in the intensive care and in the hospital
Incidence of re-intubation after surgery | From the end of surgery until 28 days after surgery
  Need to reintubate after extubation after surgery
Acute kidney injury (AKI) | From the end of surgery up to 28 days after surgery
  The definition of AKI is based on Kidney Disease; improving global outcomes (KDIGO) classification
The composite incidence of death, disabling stroke, grade 2 or 3 PGD at 72 hours, major bleeding, vascular complications, or stage II or III acute kidney injury | From the end of surgery up to 3, 14, 28 and 90 days.
  Composite outcome of potential complications related to routine and on-demand ECMO
Average financial costs and sustainability metrics | From the beginning of surgery until 28 days after surgery
  The average dollar costs and waste in kg per patient related to the use of ECMO, including perfusionist labour and all materials.
Incidence of postoperative stroke / cerebrovascular accident | From the end of surgery up to 28 days after surgery
  Stroke, disabling stroke or non-disabling stroke.
  1. Stroke: Duration of a focal or global neurological deficit ≥ 24 hours; OR &amp;lt; 24 hours if neuroimaging shows a new hemorrhage or infarct; OR the neurological deficit results in death
  2. Disabling stroke: A modified Rankin Score (mRS) of ≥ 2 at three days OR an increase in at least one mRS category from baseline for individuals with a pre-stroke baseline ≥ 1 16,17.
  3. Non-disabling stroke: An mRS score of &lt; 2 at 14 days or one that does not increase in at least one mRS category from an individuals pre-stroke baseline
Incidence of postoperative bleeding complications | From the end of surgery up to 28 days after surgery
  The definition of bleeding complication is based on Bleeding Academic Research Consortium (BARC) classification. Bleeding is defined as Major or Minor.
Duration of mechanical ventilation in hours | Beginning from the arrival to the intensive care unit immediately after surgery
  BiPAP and CPAP are not considered mechanical ventilation. Tracheostomy is not considered mechanical ventilation if a ventilator is not needed.
Incidence of postoperative tracheostomy | From the end of surgery until 28 days after surgery
  Need for a tracheostomy after surgery in a patient without a previous tracheostomy
Incidence of vascular complications | From the end of surgery to 28 days after surgery
  Major or minor vascular complications (see protocol)

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Univeristy of Alberta & Alberta Health Services, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - University Health Network / Toronto General Hospiatl, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nasir BS, Weatherald J, Ramsay T, Cypel M, Donahoe L, Durkin C, Schisler T, Nagendran J, Liberman M, Landry C, Overbeek C, Moore A, Ferraro P. Randomized trial of routine versus on-demand intraoperative extracorporeal membrane oxygenation in lung transplantation: A feasibility study. J Heart Lung Transplant. 2024 Jun;43(6):1005-1009. doi: 10.1016/j.healun.2024.02.1454. Epub 2024 Feb 28. PMID 38423414